CLINICAL TRIAL: NCT00397540
Title: Prospective Cohort Study of the Effect of Serum HBV DNA Level on Intrahepatic Recurrence in Locally Treatable, HBV-related HCC Patients
Brief Title: The Effect of Viral Load on Intrahepatic Recurrence in Hepatitis B Virus (HBV)-Related Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2006-001
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Hepatocellular; Chronic Hepatitis B
Keywords: HBV DNA; HCC; recurrence; PEIT; RFTA
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B, Chronic; Recurrence | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous ethanol injection therapy (Active Comparator): Patients with hepatocellular carcinoma who will be treated with PEIT (percutaneous ethanol injection therapy)
  Interventions: Procedure: PEIT
- radiofrequency thermal ablation (Active Comparator): Patients with hepatocellular carcinoma who will be treated with RFTA (radiofrequency thermal ablation)
  Interventions: Procedure: RFTA

INTERVENTIONS:
Procedure: PEIT — Percutaneous Ethanol Injection Therapy
  Other Names: PEI, local ablation therapy
  Arms: percutaneous ethanol injection therapy
Procedure: RFTA — Radiofrequency Thermal Ablation
  Other Names: RFA, local ablation therapy
  Arms: radiofrequency thermal ablation

SUMMARY:
The purpose of this study is to evaluate the effect of serum hepatitis B virus (HBV) DNA level on intrahepatic recurrence in locally treatable hepatocellular carcinomas (HCCs) related with HBV.

DETAILED DESCRIPTION:
Prospective cohort study

Survival

* Overall survival rate
* Disease free survival rate

Recurrence

* Cumulative recurrence rate

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* Maximal tumor size less than 5 cm
* No previous history of treatment for hepatocellular carcinoma
* Recurrent hepatocellular carcinoma located more than 2 cm from the previous cancer site and is found more than 1 year's gap

Exclusion Criteria:

* Hepatocellular carcinoma in portal vein
* Hepatocellular carcinoma in hepatic vein

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2004-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, Professor, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo JY, Kim W, Kwon JH, Jin EH, Yu SJ, Kim HY, Jung YJ, Kim D, Kim YJ, Yoon JH, Lee HS. Noninvasive fibrosis indices predict intrahepatic distant recurrence of hepatitis B-related hepatocellular carcinoma following radiofrequency ablation. Liver Int. 2013 Jul;33(6):884-93. doi: 10.1111/liv.12132. Epub 2013 Mar 5. PMID 23461618
- [Derived] Chung GE, Kim W, Lee JH, Kim YJ, Yoon JH, Lee JM, Lee JY, Kim SH, Kim D, Lee HS. Negative hepatitis B envelope antigen predicts intrahepatic recurrence in hepatitis B virus-related hepatocellular carcinoma after ablation therapy. J Gastroenterol Hepatol. 2011 Nov;26(11):1638-45. doi: 10.1111/j.1440-1746.2011.06777.x. PMID 22011297

RESULTS

PARTICIPANT FLOW:
Groups:
- Percutaneous Ethanol Injection Therapy: 99% of ethanol injected using standard percutaneous ethanol injection therapy (PEIT) intervention technique under the guidance of ultrasonography. Each procedure usually comprises 2 to 3 sessions.
- RFTA: high ultrasonic wave energy applied using standard radiofrequence thermal ablation (RFTA) intervention technique by incurring coagulation necrosis. Each procedure usually comprises only one session.
Period: Overall Study
Arm/Group | Percutaneous Ethanol Injection Therapy | RFTA
Started | 60 | 85
Completed | 59 | 85
Not Completed | 1 | 0
Not completed — short follow-up duration < 12 months | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PEIT: 99% of ethanol injected using standard percutaneous ethanol injection therapy (PEIT) intervention technique under the guidance of ultrasonography. Each procedure usually comprises 2 to 3 sessions.
- Total: Total of all reporting groups
Arm/Group | PEIT | RFTA | Total
Number analyzed (Participants) | 60 | 85 | 145
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 72] | 58 [27 to 71] | 56 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 45 | 74 | 119
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 60 | 85 | 145
Treatment modality [Number; unit: participants] | 60 | 85 | 145

OUTCOME MEASURES:

1. Primary Outcome: 1,3,5 Year-Disease Free Survival (or Recurrence Free Survival)
Description: The disease free survival is defined as the total number of surviving participants without intrahepatic recurrence of hepatocellular carcinoma for 1, 3, and 5 years.
Time Frame: 1,3,5 year
Population: ITT analysis
Measure: Number; unit: participants
Arm/Group | PEIT | RFTA
Number analyzed (Participants) | 62 | 84
participants
  1 year-disease free survival | 11 | 13
  3 year-disease free survival | 25 | 34
  5 year-disease free survival | 26 | 37

2. Secondary Outcome: Overall Survival
Description: Overall Survival: Number of Participants who Died
Time Frame: through study completion, an average of 3 years
Measure: Number; unit: participants
Arm/Group | Percutaneous Ethanol Injection Therapy | RFTA
Number analyzed (Participants) | 60 | 85
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Percutaneous Ethanol Injection Therapy | RFTA
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/85
Other Adverse Events (participants affected / at risk) | 0/60 | 0/85

LIMITATIONS AND CAVEATS:
nothing to comment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No